CLINICAL TRIAL: NCT02327494
Title: Prospective Study to Evaluate the Central Venous Oxygen Saturation and the Regional Cerebral Oxygen Saturation Monitoring at Different Stages of Neuromuscular Blockade in High-risk Patients Scheduled for Colorectal Surgery
Brief Title: Study to Evaluate Oxygen Monitoring at Different Stages of Neuromuscular Blockade in Colorectal Surgery
Acronym: OXYMUBLOC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Antoni Sabate, Professor, Hospital Universitari de Bellvitge
Other Study IDs: PR254/14
Record Dates: First submitted 2014-12-03; First posted 2014-12-30 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Colorectal Cancer
Keywords: Neuromuscular blockade; Laparoscopy; Oxygen measurements
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Neuromuscular Blockade; Rocuronium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: neuromuscular blockade — to determine the influence on oxygantion saturation parameters of the administration of neuromuscular blockade drug, rocuronio, to provide intense neuromuscular blockade during laparoscopic colorectal surgery
  Other Names: rocuronio

SUMMARY:
Anesthesia favouring deep/intense neuromuscular blockade during laparoscopy may restore hemodynamics. However, no studies has been performed comparing oxygenation parameters during laparoscopy in colorectal surgery in either moderate or intense neuromuscular blockade.

The investigators aim to investigate whether the intense neuromuscular blockade produces a better oxygenation profile measured by the central venous oxygen saturation than the moderate neuromuscular blockade.

This is a one centre, prospective clinical trial to compare oxygenation data at different stages of neuromuscular blockade in high-risk patients scheduled for colorectal surgery. Data recording will be blinded to the anesthesiologist in charge of the patient, who will manage patients by a determined protocol, based on stroke volume data to direct fluidotherapy. Data analyzer will be not be involved in the study design or in writing reports from the study. Inclusion criteria: Be a candidate to a colorectal surgical resection procedure and one of these conditions: ≥ 70 y.o, or respiratory co-morbidity, or cardiac co-morbidity or haemoglobin level < 11g/dl. The primary outcome is the absolute number of the central venous oxygen saturation, measured at the following points: basal, after tracheal intubation, before pneumoperitoneum or abdominal incision, after pneumoperitoneum or abdominal incision, 5 and 10 minutes before administration of rocuronio to produce intense blockade, continuously during profound neuromuscular blockade until the end of surgery, before sugammadex administration, after sugammadex administration, after tracheal extubation, for the 24 hours post surgical. Data of the regional cerebral oxygen saturation will be measured at the same points.

The investigators hypothesize that oxygenation data will be favourable by applying the intense neuromuscular blockade in comparison with moderate neuromuscular blockade. Also, the investigators hypothesize that oxygenation data obtained during the whole procedure including the first 24-hours post-surgery, measured by the regional cerebral oxygen saturation are comparable to data obtained by the central venous oxygen saturation. The investigators want to obtain information about influence in the outcome of producing profound neuromuscular blockade during laparoscopy colorectal by comparison of outcome data with matched historical control.

DETAILED DESCRIPTION:
The primary objective are to determine changes in the central venous oxygen saturation (ScvO2) and in the regional cerebral oxygen saturation (rSO2), measured at the following points: basal, after tracheal intubation, before pneumoperitoneum or abdominal incision, after pneumoperitoneum or abdominal incision, 5 and 10 minutes with moderate neuromuscular blockade and before administration of rocuronium to produce intense neuromuscular blockade, 5 and 10 minutes after the intense neuromuscular blockade is produced, at the end of surgery before sugammadex administration, after sugammadex administration, and after tracheal extubation.

Primary end-points:

The absolute number of ScvO2 values at the previously described points and at any fluid and drug administration related to Goal-therapy protocol

Secondary end-points:

The absolute number of rSO2 values at the previously described points and at any fluid and drug administration related to Goal-therapy protocol Any decrease of ScvO2 or rSO2 > 10% of the referee value The stroke volume value measured at same points. Plasmatic values of hemoglobin, creatinine, arterial oxygen pressure, arterial carbon dioxide pressure, Bicarbonate, pH, potassium, Sodium, glucose, lactate. Abdominal and pneumoperitoneum pressures at the previously determined points. Outcome variables and daily cost of patient

Patients, included on basis of inclusion criteria that accept to participate in the study, in whom the laparoscopy procedure starts but completed for any reason as an open procedure, will be considered as intention to treat and considered for comparison in the laparoscopy group.

Patients selected for the laparoscopy procedure, in whom the laparoscopy procedure do not start for any reason, performing instead a open procedure, will follow the study procedures and managed by the same protocol. Data of these patients will be collected and used as control group for comparison with laparoscopy group.

All outcome data collected in both laparoscopy and open procedures will compared with the outcome data of a random matched historical control group for the period 2013-2014.

Study Procedures All patients are placed in sniffing position to make mask ventilation and airway management easier. Standard monitoring (automated blood pressure cuff, electrocardiography, pulse oximetry and capnography) will start. Non-invasive Pulse determination of stroke volume (SV) monitoring (ClearSigh. Edwards) start as well as the entropy electroencephalogram monitoring (General Electric). Regional cerebral Oxygen monitoring-rSO2 (Covidien) will start at this point All patients will place on a warm blanket of convection air (Warm-Touch, Mallincrodt Medical, St. Louis, MO). After oxygen administration for 5 minutes, anesthesia induction starts which is be accomplished with 3 µg.kg-1 of fentanyl followed by 2mg.kg-1 of propofol and 0.6 mg.kg-1 of rocuronio is administered to facilitate tracheal intubation. At this point, central venous cannulation and central venous oxygen monitoring-ScvO2 (Preset Oxymetry, Edwards) starts. Sevoflurane and fentanyl will be administered to maintain entropy values <60.

Neuromuscular transmission is monitored by acceleromyography at the adductor pollicis (TOF-Watch SX; Organon Ltd. ,Dublin.Ireland), according to good clinical practice recommendation. After careful placement of appropriate electrodes and skin preparation, supramaximal stimulation is produced and the gain is adjusted to obtain a twitch height of 100% using a T1 of the Train of four (TOF mode of stimulation) as calibration, after that the initial dose of 0.6 mg.kg-1 of rocuronio is administered. Proper warm and immobilization of extremity is done. We start to recorder the monitoring of TOF stimulation at 2 Hz every 20 s. This period is considered the patient has a moderate neuromuscular blockade, defined by the reappearance of T1 on TOF stimulation. We maintain moderate neuromuscular blockade until 10 minutes after pneumoperitoneum. At this point, intense neuromuscular block (defined as no response to TOF stimulation detected in addition to no response to Post-tetanic stimulus) is produced by the administration of 0.15 mg.kg-1 of rocuronio plus a continuous infusion of 0.3 mg.kg-1.hour to maintain no response to post-tetanic count during the surgical procedure. At the end of procedure sugammadex, 4 mg. kg-1, is administered to reverse the neuromuscular blockade. Additional doses of sugammadex (2 mg.kg-1) are administered to achieve the complete reversal of neuromuscular blockade (TOF ratio > 90%), when necessary. Tracheal extubation will take place when the patient is fully awake and breathing comfortably, then patients are transferred to the surgical intensive care unit-sICU.

Intraoperative Goal Directed Therapy Protocol Management

All patient are administered a basal fluidotherapy perfusion of Ringer solution (1.5 ml/kg/h) during surgery. Steps of the Goal Directed Therapy Protocol:

* First determination of the Stroke volume (SV) is measured once the patient is placed in the OR.
* A new determination of SV is performed after the anesthesia induction and monitoring of the patients is completed, which is considered the SV referee value to optimise fluidotherapy. Afterwards, 250 ml bolus of Ringer solution is administered and a new SV is measured. If SV increases >10%, one-second bolus of 250 ml of Ringer solution is administered. The resulting stroke volume will be considered as a reference for the rest of the intervention. This determination will be considered BASELINE Stroke Volume (BSV).
* In case of the stroke volume does not increase > 10%, no additional boluses is administered, and this determination is considered BASELINE Stroke Volum (BSV).
* At any event during surgery and at the specific points the SV is measured:

If the SV remains unchanged from the baseline value (BSV), no further boluses of ringer are administered. If the actual determination of SV decreases > 10% of BSV, a bolus of 250 ml of Ringer solution is administered, and a new determination of SV is done. In case of the stroke volume increases > 10%, a second bolus of Ringer solution is administered to optimize fluid therapy. In case that SV do not increase or increase <10% of BSV, the central venous oxygen saturation (cvSO2) will be measured: If ScvO2 ≥70%, then continue to monitor stroke volume. If ScvO2 <70% check for Haemoglobin (Hb). Correction of hemoglobin <9g/dl is done by transfusion of one red cell's packed, until the target of Hb 9g/dl is achieved. If Hb is ≥ 9, then check for Cardiac index (CI): If CI ≥ 2.5 ml/min/m2, continue to monitor stroke volume. If CI < 2.5 ml/min/m2, then start Dobutamine at 2.5 mcg/Kg/minute, in a dilution of 5 mg/ml (250 mg in 50 ml), increasing the dose until the CI target is achieved.

Postoperative Goal Directed Therapy Protocol Management

* The basal fluid therapy perfusion will be 0.5 ml/kg/h of Ringer solution plus Dextrose 10% 500 ml/24 h until oral fluid administration.
* A new determination of SV is performed once the patient arrives to sICU, then a bolus of 250 ml of Ringer solution will be administered and a new SV determination is done, if it remains in the range of 10% increase change from the previous SV, it is considered the Postoperative stroke volume of reference (PSV), and no further boluses of ringer will be administered. If the actual determination of SV increases more than the 10% of value of PSV, a second bolus of 250 ml of Ringer solution will be administered, and the new SV determination will be considered the PSV.
* Repeat SV determination each 4 hours or at any event during the first 24 hour postsurgery In case of the stroke volume decreases > 10% of PSV, a bolus of ringer is administered. If the following determination of SV increases > 10% of value of PSV, a second bolus of 250 ml of Ringer's solution will be administered. In case of the stroke volume does not increase more than 10% of PSV after the bolus of ringer, the central venous oxygen saturation is measured: If ScvO2 is ≥ 70% continue monitoring stroke volume. If ScvO2 is < 70% check for Haemoglobin (Hb). If Hb is <9 g/dl, transfuse one red cell's packed. If Hb is ≥ 9 g/dl, check for Cardiac index. If CI is ≥ 2.5 l/min/m2 continue monitoring SV. If CI is < 2.5 l/min/m2 start Dobutamine at 2.5 mcg/Kg/minute, in a dilution of 5 mg/ml (250 mg in 50 ml). Increase the dose until the CI target is achieved.

Statistics For sample size calculation related to intragroup comparison at different stages of neuromuscular blockade during surgery, we consider an absolute difference of 25% of the lowest mean value, either rSO2 or ScvO2, between profound neuromuscular blockade and previous neuromuscular blockade. We consider a bilateral nonparametric-paired test, beta error of 0.2 and significance level of alfa error of 0.05. A 10% of lost patients are assumed. A total of 70 patients are considered to demonstrate differences between both neuromuscular blockades.

Is expected to have a minimum 300 determined measurement pairs. We consider 30% of pair's disagreement. A minimum of 60 patients will be recruited to perform the agreement study.

An interim analysis will be performed once 50 patients will be included in the study to demonstrated primary objective. If early benefits are achieved, the trial will be stopped. Also, trial will be stopped if the results will be inconclusive

Both, intention to treat analysis and completed cases analysis will be done. Laparoscopic reconversion to an open procedure will be treated as both: intention to treat and per protocol. Descriptive analysis will be performed using the usual measures of centrality and dispersion. Each determination of ScvO2 and rSO2 will be registered before intervention and each minute to five minutes after intervention. The worst number will be selected for analysis. The mean and standard deviation (SD) will be determined. For all comparison two-sided tests with a significance level of 5% will be used. The statistical analysis will be performed in both per protocol and intention to treat.

Primary end-point Paired data comparison:

The absolute number of rSO2 and ScvO2 values, measured during surgery and during the 24-hours period postsurgery., will be analyzed by using paired nonparametric tests (normality can be assumed or not). Paired data compared will be after each measurement with the previous.

Secondary end-points Bland-Altman representation will be used for comparison of bias and interpatient variation. ScvO2 is the goal standard, so calculation will refer to it. Definitions: Bias, averages of value differences/mean values (expressed as %); interpatient variability, 2SD of mean value; Precision, 2SD/mean value. Correlation between trend-line of both determinations also will be calculated

Intergroup Comparison, open and laparoscopic groups:

Continuous variables will be compared between using parametric test (ANOVA). Discontinuous variables will be compared using Chi-square test.

Intersample Comparison, Matched random -2013-14 historical sample:

Continuous variables will be compared with actual sample using using parametric test (ANOVA). Discontinuous variables will be compared using Chi-square test.

Cases report forms for collecting relevant variables of each patient will be created. The data is processed and stored in an electronic database for further analysis. An independent study monitor will verify the selection of cases, the existence of consent, the registration of direct and indirect complications in patients and the quality of survey data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective colorectal surgery
* With one of these following conditions: ≥ 70 year old; Respiratory co-morbidity defined as: obstructive pulmonary disease diagnosed by abnormal spirometry test, alveolar-arterial oxygen differences >15 mmHg, Sleep apnea syndrom by Eporhw criteria; Cardiac co-morbidity determined by New York functional Class II-IV; Plasmatic Hemoglobin level < 11g/dl

Exclusion Criteria:

* < 70 y.o. without respiratory or cardiac disease
* Known history of thromboembolic events in 30 days
* Known or suspected pregnancy
* Known or suspected allergy to any drug or related products used to provide anesthesia.
* Known presence of congenital disorder.
* Patients treated with aspirin, warfarin and other anti haemostatic drugs
* Contraindications to dobutamine
* Patient reluctant to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates are all adult patients (over 18 y.o) on the waiting list for elective oncologic colorectal surgical resection procedure.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
the central venous oxygen saturation (ScvO2) | intraoperative and 24 hours postoperative period
  The primary objective is to study the central venous oxygen saturation (ScvO2) measured at the following points: basal, after tracheal intubation, before pneumoperitoneun or abdominal incision, after pneumoperitoneun or abdominal incision, 5 and 10 minutes before administration of rocuronium to produce intense neuromuscular blockade, continuously during profound neuromuscular blockade until the end of surgery, before sugammadex administration, after sugammadex administration, after tracheal extubation, first 24 hour postsurgery.

SECONDARY OUTCOMES:
the central venous oxygen saturation (ScvO2)the regional cerebral oxygen saturation (rSO2) | intraoperative and 24 hours postoperative period
  Oxygen desaturation events, defined as absolute values of rSO2 below 75% or ScvO2 below 70
the regional cerebral oxygen saturation (rSO2) | intraoperative and 24 hours postoperative period
  measured at: basal, after tracheal intubation, before pneumoperitoneun or abdominal incision, after pneumoperitoneun or abdominal incision, 5 and 10 minutes before administration of rocuronium to produce profound blockade, continuously during intense neuromuscular blockade until the end of surgery, before sugammadex administration, after sugammadex administration, after tracheal extubation and at any fluid and drug administration related to Goal-therapy protocol as documented during surgery and during the 24-hours period post-surgical
Stroke volume | intraoperative and 24 hours postoperative period
  Stroke volume measured at: basal, after tracheal intubation, before pneumoperitoneun or abdominal incision, after pneumoperitoneun or abdominal incision, 5 and 10 minutes before administration of rocuronium to produce profound blockade, continuously during intense neuromuscular blockade until the end of surgery, before sugammadex administration, after sugammadex administration, after tracheal extubation and at any fluid and drug administration related to Goal-therapy protocol as documented during surgery and during the 24-hours period po
Fluidotherapy and Blood components transfusion | intraoperative and 24 hours postoperative period
  intraoperative and 24 h. postoperative fluid administration
  - Any blood product administration intraoperatively and during the first 24 h.
pneumoperitoneum and abdominal pressures | intraoperative and 24 hours postoperative period
  Abdominal pressure during intraoperative, at arrival to sICU and 24 h. postoperative in sICU
  - Pneumoperitoneum pressure minimim and maximum values
postoperative outcome | 90 days-postsurgery
  Inhospital, 30-day and 90-day postoperative mortality
  * Need for mechanical ventilation for more that 6 h. in the postoperative.
  * Cumulative hour required of mechanical ventilation at postoperative period
  * Need for reoperation
  * Re admittance to sICU
  * Need for renal replacement therapy
  * Wound infection and its graduation (superficial, deep, organ)
  * Any nosocomial infection during the hospital stage
  * Any complication related to surgical or anesthetic management, including monitoring complications, not restricted to sICU and extended to inhospital stage.
  * Changes in the postoperative Chest X-Ray not visible in the preoperative chest X-ray
  * Cost of any medical intervention related to intraoperative and postoperative patient's management
  * Cost of monitoring
  * Daily cost of patient
  * sICU and Hospital lengths of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Sabate, MD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, Barcelona, Barcelona, Spain